CLINICAL TRIAL: NCT06777459
Title: Study of Nitrate-Rich Juice on Cognitive Function in Heavy Alcohol Drinkers: a Two-Stage Adaptive Design Real-World Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Hongqiang Sun, Vice President of Peking University Sixth Hospital, Peking University Sixth Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: （2025）PKUh6（3）
Record Dates: First submitted 2025-01-07; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Heavy Drinking
Keywords: Heavy Drinking; Cognitive Function; Nitrate; Two-stage adaptive design; Real World Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RWS (Experimental): Interventions:Dietary Supplement: nitrate-rich beetroot juice
  Interventions: Dietary Supplement: Nitrate-rich beetroot juice

INTERVENTIONS:
Dietary Supplement: Nitrate-rich beetroot juice — Nitrate-rich beetroot juice, ~750 mg NO3- /d

SUMMARY:
It is known that alcohol consumption can lead to cognitive impairment and dysregulation of inflammatory responses. A preliminary randomized controlled trial conducted by our research team has suggested that nitrate may improve cognition in hospitalized patients with alcohol dependence. To further expand the population and applicability, this study aims to explore the effects of nitrate on cognition in a real-world population of heavy drinkers. The researchers have designed a two-stage clinical trial: the first stage involves the analysis of existing data, and the second stage will recruit 43-54 new participants for a 14-day dietary inorganic nitrate (nitrate-rich beetroot juice, ~750 mg NO3- /d) intervention.

DETAILED DESCRIPTION:
No comments

ELIGIBILITY:
Inclusion Criteria:

A. Individuals with a history of heavy alcohol consumption (as defined below), who have continued heavy drinking within the past week and have no plans to quit drinking within the next month.

B. Individuals with a history of heavy alcohol consumption who are currently hospitalized due to alcohol dependence or alcohol use disorder, and are still undergoing treatment.

The CDC (Centers for Disease Control and Prevention) defines heavy alcohol consumption as follows: For males: more than 15 standard alcoholic drinks per week. For females: more than 8 standard alcoholic drinks per week. Here, one standard drink unit is approximately 14 grams of pure alcohol- C. A Montreal Cognitive Assessment (MoCA) score greater than 13.

Exclusion Criteria:

A. Individuals with a history of or current infectious diseases. B. Individuals with a history of or current severe cardiovascular, cerebrovascular, hepatic, or renal diseases.

C. Individuals who are allergic to any substances used in the trial, such as beets.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of responders with a DMS-PCAD score improvement of 6 or more after intervention compared to baseline | baseline and post-intervention(two weeks after baseline test)
  Test by DMS-PCAD (Delayed Match to Sample Percent Correct , all delays) The score range is from 0% to 100%, with higher scores indicating better performance in visual memory and matching tasks.

SECONDARY OUTCOMES:
Changes of Spatial Working Memory Between Errors from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by SWM-BE (The Spatial Working Memory Between Errors ) The SWM-BE score range is primarily based on the number of errors, typically ranging from 0 to 10 errors. The higher the score, the fewer the errors, and the better the performance.
Changes of cognitive function from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by Cambridge Neuropsychological Test Automatic Battery，CANTAB
Changes of oral microbiota from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Saliva samples were used to test the composition of microbiota by 16S RNA sequencing.
Changes of inflammatory factors levels in serum from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  We collected serum sampleWs were used to test the levels of inflammatory factors by Elisa
depression | baseline and post-intervention (two weeks after baseline test)
  Test by Self-Rating Depression Scale
anxiety | baseline and post-intervention(two weeks after baseline test)
  Test by Self-Rating Anxiety Scale
Sleep Quality | baseline and post-intervention (two weeks after baseline test)
  Test by pittsburgh sleep quality index
Cognitive | baseline and post-intervention (two weeks after baseline test)
  Test by Montreal Cognitive Assessment
Dream | baseline and post-intervention (two weeks after baseline test)
  Test by Dream Evaluation Scale

IPD SHARING:
Plan to Share IPD: No